CLINICAL TRIAL: NCT06164340
Title: Retrospective Investigation of Lifestyle and Socio-cultural-economic Determinants Driving to Early Adiposity Rebound (FACILITY)
Brief Title: FACILITY: Feeding the fAmiLy: the Intergenerational approaCh to fIght obesiTY
Acronym: FACILITY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Buzzi Children's Hospital (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Valeria Calcaterra, Principal Investigator, Buzzi Children's Hospital
Other Study IDs: 03102023; CUP: F13C22001210007 (Other Grant/Funding Number: PNRR - MUR)
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Obesity, Childhood; Obesity, Maternal; Overweight
Keywords: Overweight; Obesity; Childhood obesity; Continuum of Care; Maternal health; Child Health; Policy; Food policies; Adiposity Rebound
MeSH Terms: conditions — Obesity; Pediatric Obesity; Pregnancy in Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group - Mother-child dyads: Case group: mother-child dyads (including children with overweight or obesity and early adiposity rebound).
- Control group - Mother-child dyads: Control group: mother-child dyads (including children with healthy weight).

SUMMARY:
The FACILITY STUDY is aimed at evaluating maternal and children social, cultural, economic and lifestyle-related risk factors for the development of childhood overweight, obesity and early adiposity rebound (EAR). This study consists of two phases: a cross-sectional phase and a retrospective case-control study.

DETAILED DESCRIPTION:
The FACILITY retrospective case-control study is conducted in one Italian hospital in Milan (Buzzi Children's Hospital) on children and adolescents (2-18 years old) with EAR and their mothers (≥ 18 years old). The estimated duration is 24 months.

The primary objective of the FACILITY retrospective case-control phase is to identify maternal and child lifestyle and health determinants of EAR associated with childhood obesity. The secondary objective is to identify culture-accepted early-tailored-efficiency "model to action" aligned with the Maternal, New-born, and Child Health (MNCH) continuum care approach. This "policy-model" will be based on the results of the retrospective study and on the analysis of the current scientific evidence and on the research of the global, national and local policies (city of Milan).

Participants of this study are mother-child dyads previously enrolled in the FACILITY cross-sectional study and willing to participate in the retrospective phase or newly enrolled patients from the hospital according to the eligible criteria. If eligible, variables related to the mothers and to the children will be retrospectively investigated with structured interviews and/or by consulting medical records.

For the mothers, anthropometric variables (height and weight during and after pregnancy) will be obtained from medical records, if available, or will be requested orally by structured interviews. In addition, pathological anamnesis and drug consumption during pregnancy will be evaluated with the same methodologies. Information related to pregnancy, supplements consumption during pregnancy, as well as dietary, smoking, and alcohol habits during pregnancy and breastfeeding will be assessed with structured interviews.

For the child, the nutritional status during the first 1000 days will be evaluated with the pediatric health booklet (weight, height/length, and head circumference). The type of breastfeeding and weaning characteristics will be investigated through a structured interview with the mothers. The child's dietary habits, physical activity, and motor gross achievement will be explored with the same methodologies.

ELIGIBILITY:
Inclusion criteria (CASE GROUP)

For mothers:

* Age ≥ 18 years old;
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Written and signed informed consent.

For the children/adolescent:

* Age > 2 years and < 18 years old;
* Early adiposity rebound (< 5 years of age);
* Overweight (between 2-3 Z-score) and obesity (≥ 3 Z-score) diagnosis according to the CDC growth charts.
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Mother and father/legal guardian had written and signed informed consent.

Inclusion criteria (CONTROL GROUP)

For mothers:

* Age ≥ 18 years old;
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Written and signed informed consent.

For the children/adolescent:

* Age > 2 years and < 18 years old;
* Early adiposity rebound (< 5 years of age);
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Mother and father/legal guardian had written and signed informed consent.

Exclusion criteria (CASE GROUP and CONTROL GROUP)

For the mothers:

* Mother had not written and signed informed consent;
* Inability to understand the Italian and English language.

For the children/adolescent:

* Endocrine disorders (hypothyroidism, hypercortisolism, growth hormone deficiency);
* Central nervous system damage (hypothalamic-pituitary damage because of surgery or trauma);
* Genetic diseases either monogenic (leptin deficiency, MC4R mutation) or pleiotropic genetic syndromes (Prader-Willi, Bardet-Biedl);
* Mother and father/legal guardian had not written and signed informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective study population will be a subgroup of the population previously enrolled during the cross-sectional study according to the previously identified eligibility criteria, specifically: mother-child dyads with overweight or obesity and early adiposity rebound (case) and mother-child dyads with healthy weight (control) will be enrolled. The control group will be matched to the cases selected on the basis of various factors (e.g., age, sex, race) to ensure to reduce confounding factors. New subjects will be enrolled according to the eligibility criteria of the retrospective study if the simple size is not reached.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Early adiposity rebound (EAR) | Day 1
  Child health booklet: early adiposity rebound (years) if minimum BMI occurred before 5 years of age.
Overweight and obesity | Day 1
  BMI percentile in the Center for Disease Control (CDC) growth charts (overweight: 85th-95th percentile/2-3 Z score; obesity ≥ 95th percentile/≥ 3 Z score).
Breastfeeding mode | Day 1
  Structured interview (exclusive breastfeeding, formula feeding, mixed mode).
Mode and characteristics of weaning | Day 1
  Structured interview (time of initiation, foods' introduction sequence and proposed portions, introduction or non-introduction of all food categories, difficulties experienced by the mother or the child, safety measures, proper feeding in accordance with appetite and satiety signals, typical food traditions of the maternal culture/ethnicity).
Eating habits between 1 and 2 years of age | Day 1
  Structured interview (food and beverages consumed at breakfast, lunch, dinner and snacks, meal skipping, dietary variety).
Physical activity during the first 2 years | Day 1
  Structured interview (minutes and/or hours of daily physical activity). Results will be compared with WHO guidelines.
Gross Motor Milestone Development | Day 1
  Structured interview (month when child started to walk). If age starting walking will be >18 months of age the child will be categorized as "late Motor Milestone".
Socio-demographic status for children | Day 1
  Structured interview: child age (year), race/ethnicity (Caucasian, Black, Medioriental, Asiatic, Hispanic), education level (none, elementary, middle school, high school, degree), number of people in the house, number of years in Italy.
Gestational weight gain | Day 1
  Difference between pre- and post-pregnancy weight (kg). The gestational weight gain will be compared with IOM Pregnancy Weight Guidelines.
Pregnancy characteristic | Day 1
  Structured interview: spontaneous or assisted pregnancy, pregnancy related-diseases, delivery mode (natural or caesarean), birth spacing (year).
Dietary pattern during pregnancy | Day 1
  Structured interview (adherence to particular nutritional advice, the person/expert who gave the nutritional information, dietary pattern followed, consumption of typical traditional food/dishes).
Supplements consumed during pregnancy | Day 1
  Structured interview (number and type of supplement consumed, period of assumption, who advised her to take the supplement).
Food knowledge | Day 1
  Structured interview (choose between food options to identify foods containing carbohydrates/dietary fiber, foods low in fats, foods richest in protein/calories, individual perception on the definition of a balanced diet and healthy eating, perception of a relationship between dietary pattern and health status).
Smoking habits during and after pregnancy | Day 1
  Structured interview. Smoking of traditional tobacco cigarettes (manufactured or hand-rolled cigarettes) or electronic cigarettes or heated tobacco product (HTP) products before, during, after pregnancy. Based on smoking declaration women will be categorized as follows: never smoker (i.e., never smoked), past smoker (i.e., current nonsmoker), current smoke (i.e., current user of tobacco or electronic cigarette or HTP products).
Alcohol consumption during pregnancy | Day 1
  Structured interview. Weekly consumption of alcohol units during and after pregnancy [1 alcohol unit = 12 g = small glass of red/white/rosé wine = can of double malt beer = small shot of hard liquor]; alcohol consumption history. Based on alcohol consumption declaration, women will be categorized as follows: abstainers (i.e., subjects who do not drink alcohol, zero Units of Alcohol (U.A.)), occasional drinkers (i.e., subjects who drink less than 1 U.A./week), and daily drinkers (i.e., subjects who regularly drink alcohol, more than 1 U.A./week).
Socio-demographic characteristics status for mothers | Day 1
  Structured interview. Mothers' age, marital status, race/ethnicity, nationality, education level, residence, number of people in the house, current job, number of children, number of years in Italy, household status, household income.

SECONDARY OUTCOMES:
Development of a "Model to action" policy to tackle childhood obesity | Day 1
  "policy-model" based on the results of the retrospective study

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Principal Investigator — Laboratory of Dietetics and Clinical Nutrition, Department of Public Health, Experimental and Forensic Medicine, University of Pavia, via Bassi 21, 27100 Pavia, Italy. Clinical nutrition Unit, General Medicine, ICS Maugeri IRCCS, 27100 Pavia, Italy; Valeria Calcaterra, Principal Investigator — Pediatric Department, Buzzi Children's Hospital, 20154 Milano, Italy. Department of Internal Medicine and Therapeutics, University of Pavia, 27100 Pavia, Italy.